CLINICAL TRIAL: NCT02718768
Title: A Multi Center Prospective Observational Study of Nerve Repair and Reconstruction Associated With Major Extremity Trauma
Brief Title: Study of Nerve Repair and Reconstruction Associated With Major Extremity Trauma
Acronym: Nerve
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: W81XWH-15-2-0074
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Nerve Injury(Ies)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center prospective observational study that will capture detailed information about the treatment and long term outcomes of 250 patients with PNI resulting from upper extremity trauma. The study will focus on a young adult population to include individuals ages 18-65. Patients with PNI will be recruited during the hospitalization for initial treatment of the upper extremity injury. Additional patients may be identified during clinic visits for on-going treatment of upper extremity injuries as nerve injuries evolve or upon referral from outside physicians. However, all eligible nerve injuries must be treated within 6 months of the initial upper extremity trauma. Outcomes will be assessed at 3, 6, 12, 18 and 24 months following diagnosis of the nerve injury. All assessments will take place in the clinic and will include a patient interview and a brief exam to evaluate sensory and motor function.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65
2. Sustained a peripheral nerve injury (including iatrogenic injuries and partial nerve injuries) resulting from upper extremity trauma meeting the following criteria:

   1. Involves injury or dysfunction to motor, or motor and sensory function of the axillary, radial, median, ulnar, or musculocutaneous nerve with injury localized distal to the brachial plexus cord level and proximal to the distal flexion crease of the wrist
   2. Involves a "mixed" nerve segment (i.e. involves a location of any of the above specified nerves that can be expected to have both sensory and motor axons present) but does not include sensory only distal terminations of the same nerves.
3. Receiving surgical treatment (i.e. exploration, neurolysis, repair or reconstruction, nerve or tendon transfer) within 6 months of the initial injury.

Exclusion Criteria:

1. Injuries to the brachial plexus roots, trunks, divisions and cords
2. Injuries to the nerves distal to the distal flexion crease of the wrist
3. Injuries that involve a distal extension of the parent nerve that is considered sensory only (superficial radial nerve, lateral ante brachial cutaneous nerve, etc)
4. Previous motor or sensory deficit prior to injury (e.g. resulting from trauma, stroke, muscular, neurologic, neuromuscular disorder, etc.)
5. Documented psychiatric disorder that limits ability to consent and maintain follow-up
6. Unable to speak either English or Spanish
7. Severe problems with maintaining follow up (e.g patients who are prisoners or homeless at time of injury or who are intellectually challenged without adequate family support).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 450 Patients with PNI that meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12-31 (Actual); Study Completion 2024-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Peripheral Nerve Injury (PNI) resulting from upper extremity trauma admitted across multiple trauma centers. | 2 years
Type of PNI resulting from upper extremity trauma admitted across multiple trauma centers. | 2 years
Treatment type of PNI resulting from upper extremity trauma admitted across multiple trauma centers. | 2 years
Treatment timing of PNI resulting from upper extremity trauma admitted across multiple trauma centers. | 2 years

SECONDARY OUTCOMES:
Surgical Complications | 2 years
  Surgical complications includes surgical site infections, wound dehiscence/breakdown, exposure of nerves and/or their repairs and reconstructions, breakdown of nerve repair and reconstruction, seroma/hematoma, and other local wound complications.
Pain Score | 2 years
  Self reported outcomes using the Brief Pain Inventory.
Sensory Function | 2 years
  Sensory function will be evaluated using the the touch test mono-filament hand evaluation kit.
Motor Function | 2 years
  Motor function will be evaluated using range of motion and the British Medical Research Council motor grading scale.
Global Hand Function | 2 years
  Global hand function will be measured using grip strength.
Disability | 2 years
  Self reported outcomes using the Disabilities of the Arm, Shoulder and Hand questionnaire (DASH).
Depression | 2 years
  Self reported outcomes using the Patient Health Questionnaire (PHQ-9).
Post Traumatic Stress Disorder (PTSD) | 2 years
  Self reported outcomes using the standard PTSD Checklist.
Return to Work or Duty | 2 years
  Self reported outcomes using the Work Productivity and Activity Impairment (WPAI) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jaimie Shores, MD, Principal Investigator — Johns Hopkins University; Lisa Reider, PhD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (17):
- United States (17):
  - Denver Health, Denver, Colorado
  - Ryder Trauma Center, Miami, Florida
  - Methodist Hospital, Bloomington, Indiana
  - University of Maryland Medical Center Shock Trauma Center, Baltimore, Maryland
  - The Curtis National Hand Center, Medstar Union Memorial Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - MetroHealth, Cleveland, Ohio
  - University of Oklahoma Medicine, Oklahoma City, Oklahoma
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia